CLINICAL TRIAL: NCT06877455
Title: Efficacy of Topical Methotrexate with Fractional CO2 Laser Versus Topical Methotrexate Alone in Treatment of Non Segmental Vitiligo
Brief Title: Topical Methotrexate with Fractional CO2 Laser in Treatment of Non Segmental Vitiligo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelrady Mahmoud, Resident of dermatology and venereology department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fractional laser for vitiligo
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Vitiligo
Keywords: fractional; co2 laser; vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: One side of each participant's body will receive fractional CO2 laser combined with methotrexate 1% gel, while the other side will receive topical methotrexate alone, with treatments randomized to avoid bias. The laser therapy consists of four sessions at three-week intervals using specific parameters. Participants will be followed up for six months, with assessments at baseline, during treatment, and post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- topical methotrexate with fractional CO2 laser versus topical methotrexate alone (Experimental): One side of each participant's body will receive fractional CO2 laser combined with methotrexate 1% gel, while the other side will receive topical methotrexate alone,
  Interventions: Procedure: Fractional CO2 laser assisted PDT

INTERVENTIONS:
Procedure: Fractional CO2 laser assisted PDT — One side of the body will receive fractional CO2 laser combined with methotrexate 1% gel , while the other side will receive topical methotrexate alone (or vice versa, randomized to avoid bias) for 3 months.
  Laser therapy will be performed as 4 sessions of 3 weeks interval using fractional ablative CO2 10,600 nm laser device (Daeshin Enterprise Co., Ltd. Model: Multixel, Seoul, Korea). A single pass will be performed at the following parameters: pulse energy 42-45 mJ, density of 100 spots/cm2 depth level of 1-2 covering an area of 1 cm2 MTX gel will be prepared in the Department of Pharmaceutics at Assiut University Patients will be followed up for total 6 months (e.g., baseline, weeks 3, 6,9,12,15 and post-treatment at months 4 and 6).

SUMMARY:
This prospective, within subject clinical trial aims to evaluate the efficacy of combining fractional CO2 laser with topical methotrexate versus topical methotrexate alone in treating non-segmental vitiligo. Patients with comparable lesions on both sides of their body will receive both treatments randomly assigned to each side. The study assesses repigmentation, safety, patient satisfaction, and quality of life over six months.

DETAILED DESCRIPTION:
The study is a prospective, within subject, self-controlled, randomized clinical trial conducted at the Department of Dermatology, Assiut University. Participants are patients aged 18-65 with stable non-segmental vitiligo, having comparable lesions on both sides of their body. They must not have received corticosteroid or phototherapy treatments in the last three months and must provide informed consent. Exclusion criteria include other skin diseases, pregnancy, severe organ dysfunction, compromised immune function, and skin type 1 with phototherapy allergy.

Intervention and Follow-Up One side of each participant's body will receive fractional CO2 laser combined with methotrexate 1% gel, while the other side will receive topical methotrexate alone, with treatments randomized to avoid bias. The laser therapy consists of four sessions at three-week intervals using specific parameters. Participants will be followed up for six months, with assessments at baseline, during treatment, and post-treatment.

Outcome Measures The primary outcome is the percentage of repigmentation, assessed through standardized digital photographs evaluated by blinded dermatologists. Secondary outcomes include safety evaluation, patient satisfaction, the pattern of repigmentation, the Vitiligo Area Scoring Index (VASI) score, and quality of life measured using a validated questionnaire.

Methods for Evaluation Photographs will be taken under Wood's lamp examination at baseline, before each treatment session, and two months after the final treatment. The efficacy will be evaluated by comparing pre- and post-treatment photographs. Safety and patient satisfaction will be assessed throughout the study period. The study aims to provide evidence on the effectiveness of combining fractional CO2 laser with topical methotrexate for vitiligo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants are patients aged 18-65 with stable non-segmental vitiligo, having comparable lesions on both sides of their body. They must not have received corticosteroid or phototherapy treatments in the last three months and must provide informed consent.

Exclusion Criteria:

* Exclusion criteria include other skin diseases, pregnancy, severe organ dysfunction, compro

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
percentage of repigmentation | 6months
  percentage of repigmentation, assessed through standardized digital photographs evaluated by blinded dermatologists

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelmaksoud A, Dave DD, Lotti T, Vestita M. Topical methotrexate 1% gel for treatment of vitiligo: A case report and review of the literature. Dermatol Ther. 2019 Sep;32(5):e13013. doi: 10.1111/dth.13013. Epub 2019 Jul 16. PMID 31265164